CLINICAL TRIAL: NCT01825551
Title: The Effect of Granulocyte Colony Stimulating Factor (GCSF) in the Treatment of Amyotrophic Lateral Sclerosis (ALS) Patients Referred to Tehran Imam Khomeini and Shariati Hospital Centers in 2013
Brief Title: The Effect of GCSF in the Treatment of ALS Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91-01-54-17265
Record Dates: First submitted 2013-03-13; First posted 2013-04-05 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Granulocyte Colony Stimulating Factor
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Granulocyte Colony Stimulating Factor (Active Comparator): Granulocyte Colony Stimulating Factor 10 microgram/ kg/ day for 5 days subcutaneously
  Interventions: Drug: Granulocyte Colony Stimulating Factor
- Placebo (Placebo Comparator): normal saline 0.01 ml/kg/day for 5 days subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor
  Arms: Granulocyte Colony Stimulating Factor
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effect off Granulocyte Colony Stimulating Factor (GCSF) in the treatment of Amyotrophic Lateral Sclerosis (ALS) patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 85
* definite or probable ALS according to revised El Escorial criteria
* maximum 2 years from initiation of symptoms to study entry
* mild to moderate disability according to revised ALS functional rating scale (ALSFRS-r)

Exclusion Criteria:

* familial ALS
* pregnancy or lactation
* myeloproliferative or hematologic disorders
* active immunological disease
* liver or renal or heart disease
* HIV positive
* significant cognitive disorder
* hypersensitivity to GCSF

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
patient's function | one year
  based on revised ALS Functional Rating scale (ALSFRS-r)

SECONDARY OUTCOMES:
mobilizing bone marrow stem cells | 1 year
  based on cluster of differentiation 34 (CD34) and white blood cell (WBC) counting
amplitude of compound muscle action potential in ulnar and peroneal nerve | 1 year
  based on compound muscle action potential (CMAP) measured in nerve conduction study
quality of life | 1 year
  based on Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ40)
muscle power | 1 year
  based on Muscle Manual Test (MMT)

CONTACTS AND LOCATIONS:
Locations (1):
- Iranian Neurology Research Center of Tehran University of Medical Sciences, Tehran, Tehran Province, Iran